CLINICAL TRIAL: NCT02200900
Title: Study of Nasopharyngeal Pressures, Tidal Breathing Indices and Inspired Gas Concentrations During High Flow Nasal Cannula (HFNC) and CPAP Treatment in Neonates
Brief Title: Study of Respiratory Physiology During High Flow Nasal Cannula Treatment in Preterm Neonates.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 7022
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Extreme Prematurity - Less Than 28 Weeks; Respiratory Distress Syndrome in Premature Infants
Keywords: High flow nasal cannula; Continuous Positive Airway Pressure; Respiratory physiology
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants | interventions — Blood Gas Monitoring, Transcutaneous; Tidal Volume

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 ( CPAP followed by HFNC) (Active Comparator): In this group pharyngeal pressure, transcutaneous carbon dioxide concentration, tidal volumes and pharyngeal gas concentrations will be recorded on CPAP first followed by HFNC.
  Interventions: Other: Pharyngeal pressure; Other: Transcutaneous carbon dioxide; Other: Pharyngeal gas concentrations; Other: Tidal volume
- Group 2 (HFNC followed by CPAP) (Active Comparator): In this group pharyngeal pressure, transcutaneous carbon dioxide concentration, tidal volumes and pharyngeal gas concentrations will be recorded on HFNC first followed by CPAP.
  Interventions: Other: Pharyngeal pressure; Other: Transcutaneous carbon dioxide; Other: Pharyngeal gas concentrations; Other: Tidal volume

INTERVENTIONS:
Other: Pharyngeal pressure — Babies will have pharyngeal pressures measured during the CPAP and HFNC respiratory support.
Other: Transcutaneous carbon dioxide — Babies will have transcutaneous carbon dioxide measured during CPAP and HFNC respiratory support.
Other: Pharyngeal gas concentrations — Measurement of pharyngeal oxygen and carbon dioxide concentration will be done during CPAP and HFNC respiratory support.
Other: Tidal volume — Tidal breathing indices including tidal volume and FRC base line changes will be recorded during CPAP and HFNC respiratory support.

SUMMARY:
The most commonly used noninvasive respiratory support in preterm babies is Continuous Positive Airway Pressure (CPAP), which provides extra breathing support to babies who are breathing by themselves). Increasingly High flow Nasal Cannula (HFNC, newer form of extra breathing support) therapy has found its way in clinical practice despite lack of good physiological data. There are also concerns about its potential to generate higher pressures in airways which can cause over distension of lungs.

We would like to find out the effects of HFNC on

* 1. Airway pressures in various flow rates and in comparison to CPAP.
* 2. Breathing markers including respiratory rate (speed of breathing), oxygen and carbon dioxide levels, tidal volumes (how much air breathed in with each breath) and airway wash out (wash out of waste gas from the airway).

We plan to study 15 babies each in three different weight categories supported with either CPAP or HFNC. The airway pressures, oxygen and carbon dioxide concentration in airway are measured by a small plastic catheter (similar to feeding tube but much shorter in length), carbon dioxide levels by skin sensors, how fast and how much babies breathe by a special vest applied like a layer of clothing. These will be recorded both on HFNC and CPAP. There are no blood tests or invasive procedures involved. The baby will be monitored throughout the study period of approximately two hours by experienced registrar who is trained to use the study device.

This study will improve our understanding of physiological effects of HFNC and lead to better care of preterm babies.

DETAILED DESCRIPTION:
Purpose and design

Design: Prospective randomised crossover study.

Purpose:

* Raising airway pressure is one of the most important interventions at the disposal of clinicians treating patients with respiratory failure. In premature infants Continuous Positive Airway Pressure (CPAP) and High Flow Nasal Cannula (HFNC) are noninvasive techniques to raise mean airway pressure when intubation is not required. It is not clear how clinicians choose between these techniques and there is little data comparing the physiological effect of these treatments.
* A composite physiological assessment of babies on HFNC and CPAP treatment is required to understand how HFNC works. It is important to answer this question to understand how best to use HFNC in babies.
* This proposal is designed to provide information on physiological effects of both therapies in same population of babies across different weight categories. The study protocol involves use of same HFNC device that is currently being used in neonatal unit.

Interventions:

1. A small plastic catheter tip transducer (Gaeltec) will be placed in upper breathing passage (nasopharynx or oropharynx) using standard methods. From this we will measure airway pressures and respiratory gas concentrations.

The catheter will be removed soon after the study is completed. This procedure will be done once during the study.

2. Breathing markers (Tidal breathing indices) will be measured by non invasive method using Volusense method where a vest will be applied over the chest and abdomen like a layer of clothing. The Volusense vest will be removed soon after the procedure. This process is done once during the study.

3. Blood carbon dioxide (CO2) levels will be measured by a non invasive transcutaneous sensor applied to the skin (Tosca Radiometer). This skin sensor will be removed soon after the study is completed.

1. The baby must be clinically stable for preceding 12 hours on noninvasive breathing support (not meeting exit criteria). The babies will be randomised to either group 1 (CPAP first followed by HFNC) or group 2 (HFNC first followed by CPAP) by computerised software programme.
2. The measuring devices namely nasopharyngeal catheter, Volusense vest and transcutaneous CO2 sensor are placed as per standard methods.
3. After ensuring babies' clinical stability the measurements are recorded at HFNC gas flow rate range from 2 litres to 8 litres per minute and in CPAP of 6 cm of water pressure level.
4. The study lasts about 2 hours. The baby spends 10 minutes at each HFNC flow rate level and 30 minutes of equilibration period when support will be changed between HFNC and CPAP.
5. Routine measurement of heart rate, respiratory rate and oxygen saturations will be done as per standard neonatal practice. The above data will be recorded electronically for analysis with total study duration around 120 minutes.
6. Respiratory support can be terminated at any point if clinically not indicated.

The researcher is an experienced neonatal registrar who will be directly observing the baby throughout the study.

Measurements would be discontinued if any pre set exit criteria is noted.

Statistics: A total of 45 babies (15 babies in each weight category: <1000 grams, 1001500 grams and >1500 grams) will be studied.

ELIGIBILITY:
Inclusion Criteria:

* They are less than 37 weeks' gestation at birth and more than 5 days of age
* Are on non-invasive respiratory support and
* The parent(s) have given written informed consent to their baby's participation

Exclusion Criteria:

* Infants who are clinically unstable and unsuitable for non-invasive respiratory support as judged by attending neonatology consultant clinician.
* Participation in a concurrent study that prohibits inclusion in other trials
* Known major upper airway, lower respiratory tract, cardiac or gastrointestinal tract anomaly
* Current complications such as pneumothorax.

Ages: 5 Days to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Nasopharyngeal pressures (pressures in upper breathing passages) generated by HFNC at flow rate range of 2 to 8 L/min. | Primary outcome recorded during the measurement period of 2 hours.
  The range of pressures generated during high flow nasal cannula treatment over flow rate range of 2 to 8 litres per minute will be recorded during the study period.

SECONDARY OUTCOMES:
Nasopharyngeal pressures (pressures in upper breathing passages) generated at CPAP of 6 cm of water | Pressures recorded during the study period of 2 hours
  The nasopharyngeal pressures recorded during CPAP of 6 cm of water pressure will be documented.
The effect of changing flow rate of HFNC on following physiological parameters Oxygen saturation and transcutaneous CO2, Respiratory rate, Tidal volume and FRC baseline change. | Recorded during the study period of 2 hours
  The physiological parameters including oxygen saturation and transcutaneous CO2, Respiratory rate, Tidal volume and Functional Residual Capacity (FRC) baseline change will be recorded by monitors during the study period.
The relationship of flow and inspired oxygen concentration on actual laryngeal inspired and expired O2 and CO2 concentration in HFNC and CPAP. | Recorded during the 2 hour study period
  The relationship of flow and inspired oxygen concentration on actual pharyngeal inspired and expired O2 and CO2 concentration in HFNC and CPAP will be noted by gas analyser.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher O'Brien, MRCP, FRCPCH, Principal Investigator — The Newcastle upon Tyne Hospitals NHS Foundation NHS Trust
Locations (1):
- The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Tyne and Wear, United Kingdom